CLINICAL TRIAL: NCT00018642
Title: Predicting the Optimal Pharmacotherapy for Outpatients With Schizophrenia
Brief Title: Quetiapine vs Haloperidol Decanoate for the Long Term Treatment of Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: MHBS-042-96F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: quetiapine; haloperidol decanoate
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate; haloperidol decanoate

INTERVENTIONS:
Drug: quetiapine
Drug: haloperidol decanoate

SUMMARY:
The purpose of this research study is to determine whether a new drug for schizophrenia is better for the maintenance treatment than a standard drugs currently prescribed. The new medication is called quetiapine and it will be compared with a standard medication called haloperidol decanoate. The study will determine if quetiapine causes fewer problems than haloperidol with side effects such as stiffness and restlessness and whether it costs the VA more or less to treat patients with quetiapine. In addition, blood samples will be collected every three months to determine if certain chemicals in the blood can influence the outcome of the subjects' illness.

ELIGIBILITY:
Inclusion Criteria

1. Schizophrenia or Schizoaffective Disorder diagnosed by DSM-IV
2. Between the ages 18-60.
3. A candidate for maintenance antipsychotic therapy. This means that patients will have had at least two documented episodes of acute schizophrenic illness or at least two years of continuing psychotic symptoms.

Exclusion Criteria

1. Organic brain disease.
2. Mental Retardation
3. Chronic medical illness which would make antipsychotic medication inappropriate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1997-04; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States